CLINICAL TRIAL: NCT01743534
Title: Impact of the Shape of Plates on the Conservation of Praxis in the Food at the Old Persons Suffering From Severe Insanities of Chap Alzheimer or Mixed in Institution.
Brief Title: Conservation of Praxis in the Food and Alzheimer Disease
Acronym: PRAXALIM
Status: Completed | Type: Observational
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Other Study IDs: I09023
Record Dates: First submitted 2011-05-30; First posted 2012-12-06 (Estimated); Last update posted 2016-08-22 (Estimated); Status verified 2011-05

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Conservation of praxies and form plates

SUMMARY:
The insanities, priority of public health in 2008, have significant prevalency in Limousin, region in the ageing demography (1/3 of the population is more than 60 years old against 1/5th of average in France). To prevent the lack of therapeutic solutions, for these evolutionary diseases, the new plan Alzheimer 2008-2012 encourages the research.

The insanities deprive gradually the individual of their autonomy, their personality and their identity. The help of an institution is sometimes inevitable. In the middle of this stressful environment, the patient affected by severe insanity, need marks.

The aspect of their old objects, significant for them, has to be prioritized because the institutional universe, often depersonalized doesn't mean anything for them. In front of repeated failures, they're hurt in their self respect.

The prevention of the undernutrition, comes by a preservation of praxis and pleasure at table. The institutional plate used in certain hospital sectors, is unpersonal (rectangular, divided) and can be destabilizing for the mentally ill person.

ELIGIBILITY:
Inclusion Criteria:

* Men and women of more than 75 years
* Patients suffering from insanities of type Alzheimer
* Severe stage of the disease
* Residents in a Hospital for dependent old persons, with its own dining room
* Persons accommodated in the clinical service for more than 30 days
* EBS score <16
* Information in the participation of the resident, their legal representative and their family
* Patients affiliated to the Social Security.
* Filled and signed form of participation
* Patient having a appointed reliable person or one helping known whose references are indicated in the patient file.

Exclusion Criteria:

* Patients presenting pathologies being able to interfere with the evaluation
* Participating patients in another research for type clinical trial.
* Undernutrition patients
* Patients presenting oral hurts
* Protected patient or having nobody helping.

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patient achieves of the Alzheimer's disease
Sampling Method: Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2011-07; Primary Completion 2016-02 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Score of Blandford Scale | 2 days
  Blandford Scale of which will be estimated before ( J0) and after ( J21) modification of the plate

SECONDARY OUTCOMES:
Score of Blandford scale | 2 days
  Blandford scale which will be estimated before ( J0) and after ( J42) modification of the plate

CONTACTS AND LOCATIONS:
Locations (1):
- Limoges University hospital, Limoges, France